CLINICAL TRIAL: NCT07210788
Title: Evaluation of Crowning Time on the Incidence of Levator Ani Muscle Avulsion
Brief Title: The Effect of Crowning Time on Levator Ani Muscle Avulsion
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Clinical Professor, Université de Sherbrooke
Other Study IDs: 2024-5391
Record Dates: First submitted 2025-08-19; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Time of the Crowning of the Fetal Head; Levator Ani Avulsion; Labor Delivery; Postpartum
Keywords: levator ani; levator ani avulsion; crowning time; crowning time of the fetal head; primiparous; singleton foetus; vertex position; postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primiparous women with singleton vertex position having a spontaneous vaginal birth: This cohort study follows primiparous women having had an unassisted by forceps or vacuum labor in post-partum with a 4D ultrasound of the perineum.

SUMMARY:
Levator ani muscle is one of the main components of perineal muscles and plays a crucial role in urinary continence and pelvic organ support. An avulsion, detachment from its insertion, of this muscle can occur during vaginal birth. It is well known that this major injury can cause many symptoms such as urinary incontinence and pelvic organ prolapses. Some risk factors of this important injury have been identified in the literature, such as the use of forceps. However, to date, no study has evaluated the impact of the crowning of the fetal head during labor on perineal muscles, specifically the levator ani muscle avulsion. Hence, the objectives of this study are to evaluate the association i) the time of the crowning of the fetal head during labor and levator ani muscle avulsion, ii) the time of the crowning of the fetal head and urogynecological symptoms, and iii) use of episiotomy and levator ani muscle avulsion. Postpartum primiparous women will undergo a 4D transperineal ultrasound to evaluate their pelvic muscles and complete questionnaires assessing urogynecological symptoms.

DETAILED DESCRIPTION:
This is a prospective cohort study evaluating the impact of the crowning time of the fetal head in the second stage of labor on the incidence of levator ani muscle avulsion. Levator ani muscle is hypothesized to avulse during the distension of the pelvic floor muscles, as during a forceps use, and most probably during the crowning of the fetal head. In the study center, the crowning of the fetal head is systematically calculated during labor by nurses and doctors. To eliminate some potential confounding factors, only primiparous women with spontaneous vaginal delivery of a vertex position baby will be recruited in the post-partum period. In order to evaluate the presence of levator ani muscle avulsion, they will be assessed with a 4D transperineal ultrasound by using a standard diagnosis protocol. The delivery hospital file will then be examined to collect potential confounding variables. Prior to data collection, all study participants will give their written informed consent. This study will add more literature to the prevention of the levator ani muscle avulsion and its long-term complications.

ELIGIBILITY:
Inclusion Criteria:

Primiparous women GxT1 At term: ≥ 37+0 weeks of gestation (included) Spontaneous vaginal delivery (SVD) Cephalic presentation History of miscarriage before 20 weeks or with a fetal weight < 350g

Exclusion Criteria:

Contraindications to vaginal delivery Assisted vaginal delivery Age under 18 years Shoulder dystocia Extensive pelvic reconstructive surgery (e.g., bladder exstrophy repair) Term intrauterine fetal demise Twin or multifetal pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population will recruit primiparous postpartum women who meet the inclusion criteria and gave birth at CHUS Fleurimont during the recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete and partial unilateral or bilateral avulsion of the levator ani muscles in the post-partum period | In the post-partum period, up to 1 year post-partum
  Diagnostic established with standard levator-urethra gap measures assessed with a transperineal 4D ultrasound
Crowning time of the fetal head | The data was obtained from the medical records of each participant during labor.
  The time between the crowning of the fetal head and birth is systematically recorded during labor at the study center for all deliveries. Only participants who meet the inclusion criteria are considered for the study.

SECONDARY OUTCOMES:
Rate and type of perineal tears | The data was obtained from the medical records of each participant during labor.
  Grade of perineal tear collected in the medical file
Incidence and severity of urogynecological symptoms | In the post-partum period, up to 1 year post-partum
  Validated questionnaires on urogynecological symptoms: PFDI-46 and ICIQ-IU-SF
  PFDI-46 (Pelvic Floor Distress Inventory - 46 Items) Full title: Pelvic Floor Distress Inventory
  Structure & Scoring: It comprises three subscales:
  1. UDI (Urinary Distress Inventory): range 0-300
  2. POPDI (Pelvic Organ Prolapse Distress Inventory): range 0-300
  3. CRADI (Colorectal-Anal Distress Inventory): range 0-400 Interpretation: Higher scores indicate worse symptom distress-i.e., a higher burden of pelvic floor symptom
  ICIQ-UI-SF (International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form) Full title: International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form Scoring: Total score: 0-21 (sum of items 3, 4, and 5; items 1, 2 are demographic, one item is unscored) Interpretation: A higher score indicates greater severity of urinary incontinence and a greater negative impact on quality of life
Use of episiotomy | The data was obtained from the medical records of each participant during labor.
  Type and use of episiotomy collected in the medical file

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Morin, PT, Study Director — Université de Sherbrooke
Locations (1):
- CHUS Fleurimont, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon approval by the principal investigator and study team.